CLINICAL TRIAL: NCT02068625
Title: Rasagiline (Azilect) - Neuroprotection for Macula-off Retinal Detachment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Persisting recruitment difficulties
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 178/10; 2012DR2022 (Other: Swissmedic)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Retinal Detachment
Keywords: retinal detachment; rasagiline; optical coherence tomography; visual acuity; neuroprotection; azilect
MeSH Terms: conditions — Retinal Detachment | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Patients getting perioperative oral treatment with rasagiline (1mg daily) for 7 days
  Interventions: Drug: Rasagiline
- Control (Placebo Comparator): Patients getting perioperative oral treatment with placebo for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rasagiline — Rasagiline 1mg daily orally for 7 days
  Arms: Treatment
Drug: Placebo — Oral treatment with placebo for 7 days
  Arms: Control

SUMMARY:
This randomised, double-blind, placebo-controlled clinical trial investigates the neuroprotective effect of rasagiline in patients suffering from a retinal detachment affecting central vision. Based on results from a study in mice suffering from retinal degeneration, the investigators hypothesize that rasagiline delays neurodegeneration in the retina and improves visual acuity outcomes after retinal detachment surgery. Rasagiline is a second-generation propargylamine with neuroprotective properties modulating the caspase-dependent pathway of programmed cell death.

DETAILED DESCRIPTION:
Background

In previous experimental studies neuroprotection by rasagiline has been shown in rds-mice, a model for slow retinal degeneration. It is known from these experiments that rasagiline specifically delays apoptosis, but also modifies inflammation and autophagy. The bioavailability of the drug in the central nervous system is high, and based on the literature is sufficient in the retina.

In retinal detachments the outer layers of the neurosensory retina are deprived of nutrients and degeneration of the photoreceptors occurs fast. This is particularly relevant in the macular area of the retina where the density of photoreceptors is high, such that visual acuity recovery can be significantly limited by photoreceptor loss.

Objective

To assess the neuroprotective effect of oral rasagiline (1mg daily for 7 days) administered perioperatively in patients undergoing surgical retinal detachment repair for central vision involving retinal detachments.

Methods

In this clinical trial, patients suffering from retinal detachments affecting the fovea get randomly assigned to perioperative oral treatment with either rasagiline (1mg) or placebo once daily for 7 days. Pharmacologic treatment is initiated at the time of hospital admission, usually the day before surgery. The main outcome of the study is visual acuity six months after surgical retinal detachment repair. Structural differences of the neurosensory retina between groups will be analysed by optical coherence tomography, a non-invasive imaging method for retinal pathology.

ELIGIBILITY:
Inclusion Criteria:

* Rhegmatogenous retinal detachment
* Central vision affected for less than 72 hours
* Pseudophakic
* Age 18 or over
* Not participating in other clinical trials
* Willing to attend follow-up visits
* Written informed consent

Exclusion Criteria

* Phakic
* Narrow angle glaucoma
* Previous intraocular surgery other than cataract operation
* Retinal disease
* Concurrent treatment with MAO inhibitors
* Pregnancy
* Malignant arterial hypertension
* Liver or kidney failure
* Life-threatening or malignant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ETDRS Visual Acuity | 6 months

SECONDARY OUTCOMES:
Central retinal thickness | 6 months
  Measured by Optical Coherence Tomography (OCT)
Number of patients with side effects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, Study Chair — Department of Ophthalmology, Bern University Hospital; Andreas Ebneter, Principal Investigator — Department of Ophthalmology, Bern University Hospital
Locations (1):
- Department of Ophthalmology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Eigeldinger-Berthou S, Meier C, Zulliger R, Lecaude S, Enzmann V, Sarra GM. Rasagiline interferes with neurodegeneration in the Prph2/rds mouse. Retina. 2012 Mar;32(3):617-28. doi: 10.1097/IAE.0b013e31821e2070. PMID 21878836
- [Background] Youdim MB, Bar Am O, Yogev-Falach M, Weinreb O, Maruyama W, Naoi M, Amit T. Rasagiline: neurodegeneration, neuroprotection, and mitochondrial permeability transition. J Neurosci Res. 2005 Jan 1-15;79(1-2):172-9. doi: 10.1002/jnr.20350. PMID 15573406
- [Background] Travis GH. Mechanisms of cell death in the inherited retinal degenerations. Am J Hum Genet. 1998 Mar;62(3):503-8. doi: 10.1086/301772. No abstract available. PMID 9497269
- [Background] Cook B, Lewis GP, Fisher SK, Adler R. Apoptotic photoreceptor degeneration in experimental retinal detachment. Invest Ophthalmol Vis Sci. 1995 May;36(6):990-6. PMID 7730033
- [Background] Eliash S, Shteter N, Eilam R. Neuroprotective effect of rasagiline, a monoamine oxidase-B inhibitor, on spontaneous cell degeneration in a rat model. J Neural Transm (Vienna). 2005 Aug;112(8):991-1003. doi: 10.1007/s00702-004-0254-4. Epub 2005 Mar 15. PMID 15765264